CLINICAL TRIAL: NCT06565728
Title: Comparative Study of the Role of Vitamin D Supplementation, Versus Sildenafil Citrate in Patients Diagnosed With Fetal Growth Restriction, Randomized Control Trial
Brief Title: Vitamin D Versus Sildenafil Citrate in Fetal Growth Restriction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Ramadan, Resident of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fetal Growth Restriction
Record Dates: First submitted 2024-07-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2022-11

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate; acetylsalicylic acid lysinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Vitamin D3 group (Active Comparator): Consists of 33 pregnant women who received oral vitamin D3 (vitamin D-3 2000 IU) and low dose aspirin.
  Interventions: Drug: Vitamin D3 2000 UNT Oral Tablet
- Group A: Sildenafil group (Active Comparator): Consists of 33 pregnant women who received oral sildenafil citrate 20 mg (Respatio) and low dose aspirin
  Interventions: Drug: Vitamin D3 2000 UNT Oral Tablet
- Group A: Control group (Active Comparator): Consists of 33 pregnant women who received low dose aspirin only
  Interventions: Drug: Vitamin D3 2000 UNT Oral Tablet

INTERVENTIONS:
Drug: Vitamin D3 2000 UNT Oral Tablet — To assess the role of vitamin D3, versus sildenafil citrate, versus control group in pregnancies complicated by fetal growth restriction
  Other Names: Sildenafil Citrate; Asprin

SUMMARY:
Fetal growth restriction, also named Intrauterine growth restriction is a prevalent disease in pregnancy , it is a descriptive term for a pathological process, and can be described as the process where a fetus who has a certain growth potential based on genetic criteria is limited in its growth because of a pathological environmental influence

DETAILED DESCRIPTION:
Fetal or Intrauterine growth restriction, describes a pathological condition in which the fetus fails to grow to its biological potential, because of poor placental function , both American society of obstetrics and gynecology of and Royal college of obstetrics and gynecology have adopted the definition of Intrauterine growth restriction as estimated fetal weight is less than 10th percentile .

It is a multifaceted problem that increases the risk of hypoxemia, acidemia, preterm deaths, and maternal distress, and disposes the infant to a number of metabolic disorders, polycythemia, lung problems, intraventricular hemorrhage, cognitive dysfunction, and cerebral palsy, which occur in both term and preterm infants .

Vitamin D deficiency is highly prevalent among pregnant women, not only vitamin D deficiency during pregnancy causes maternal and fetal side effects, it also increases the risk of preeclampsia, gestational diabetes, preterm birth, and birth of a child younger than small for gestational age, inadequate fetal immune system, wheezing and eczema, and risk of respiratory infections in the infants.

Vitamin D is a transcriptional regulator of endothelial NO synthase, effectively increasing the production of NO, the most potent vasodilator within the vasculature. previous Studies showed that the vitamin-D receptors play a critical role in maintaining vascular health, and this assumption was supported by data Showing reduced NO production.

It was suggested that vitamin D improves vascular function via reducing the production of NO-scavenging oxygen radicals and subsequently improving NO bioavailability and maintain vascular health.

Vitamin D level during the pregnancy in women with low-birth-weight infants was significantly lower than its level in other women. It was eventually found that vitamin D level in pregnancy was effective in bone metabolism and growth process of the fetus .

Vitamin D deficiency during pregnancy causes potentially harmful implications in the mother and the fetus. Several studies have referred to the relationship between vitamin D deficiency and the incidence of intrauterine growth retardation.

Some studies have shown that increasing the amount of 25-hydroxy vitamin D in the bloodstream before and during pregnancy contributes to nesting and causes stability in pregnancy, as well as increased calcium uptake required for fetal growth and development.

Studies have also indicated that the decreased expression of vitamin D receptors results in functional impairment and limitation in the beneficial effects of vitamin D in regulating the fetus-placental growth.

Maternal vitamin D deficiency was observed in all pathological pregnancies with a decrease in the staining levels of placental vitamin D receptor in intrauterine growth retardation. And severe vitamin D deficiency may play an important role in placental inflammation, which in turn may lead to a higher risk of intrauterine growth retardation and other neonatal side effects.

Vitamin D supplementation doses should be: 1500-2000 IU/day, necessary for maintaining 25(OH)D serum level above 30 ng/mL, currently available studies seem to recommend starting prophylaxis with vitamin D at the beginning of the pregnancy, to be continued throughout the entire pregnancy and during lactation.

The standard options for management of intrauterine growth retardation are expectant management till pregnancy termination. This involves modification of maternal lifestyle together with fetal surveillance, since impaired placental circulation is a major cause, vasodilators may have their role .

Sildenafil citrate (trade name: Revatio, Viagra, Respatio, etc.) was emerged as a drug helping vasodilation which may represent an effective intervention for intrauterine growth retardation pregnancies with dose of 20 mg once daily. Studies showed that mean birth weight at delivery was increased significantly with sildenafil usage. Of course, this had its value in decreasing admission to the newborn nursery unit.

Sildenafil citrate treatment may present a new hope towards better perinatal outcomes for pregnancies complicated by intrauterine growth retardation that may help to decrease neonatal admission to newborn nursery.

Sildenafil citrate induces vasodilation through inhibition of type 5 phosphodiesterase (PDE5) which is responsible for the degradation of cGMP to guanosine monophosphate. Therefore, inhibiting PDE5 delays the breakdown of cGMP and increases vasodilation.

ELIGIBILITY:
Inclusion Criteria:

1. Women with singleton spontaneous pregnancy with fetal growth restriction more than 28 weeks, confirmed by ultrasound based on estimated fetal weight and measurement of abdominal circumference (AC)< 10th percentile for gestational age or lag of two weeks or more between the current measurements and expected one, dating since the first trimester of pregnancy.
2. Age 20- 40 years.
3. Patients with regular menstrual pattern before pregnancy.
4. Patients are able to attend follow up as planned.

Exclusion Criteria:

1. Patients with uncertain gestational age
2. Maternal cardiovascular disease (congenital, ischemic and rheumatic heart diseases), diabetes, kidney disease, hepatic disease, anemia, antepartum hemorrhage and placenta previa.
3. Patients with known or suspected foetal anomalies
4. Fetal growth restriction because of severe preeclampsia.
5. Use of vasodilator medication.
6. Multiple pregnancies
7. Smoking, drugs or alcohol abusers.
8. Obstetric complications (intrauterine infection, bleeding, premature rupture of membranes).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Gestational age Measurements | 6 months
  Estimation of The Gestational age at the week 28 of gestation by measuring fetal head circumference, Abdominal Circumference and fetal femur length.

CONTACTS AND LOCATIONS:
Overall Officials: Omneya Mostafa Helal, Professor, Study Chair — Department of Obstetrics and gynecology. Faculty of Medicine, Cairo University; Marwa Mohamed Mahmoud Eid, M.D, Study Director — Department of Obstetrics and gynecology. Faculty of Medicine, Cairo University
Locations (1):
- kasr Alainy University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No